CLINICAL TRIAL: NCT01257854
Title: Polymorphisms and Busulfan Pharmacokinetic Study in Pediatric Transplnatation
Brief Title: Polymorphisms and Busulfan Pharmacokinetic Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Principal Investigator, Marc Ansari, MD, PhD, University Hospital, Geneva
Other Study IDs: 2009-018105-41; 2009-018105-41 (EudraCT Number)
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Children Who Receive a Stem Cell Transplantation With Busulfan IV
Keywords: busulfan; pharmacogenetic; pharmacokinetic; toxicity; survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA from each patient are kept. Plasma from some centers are kept
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Busulfan, pharmacogenetic, pharmacokinetic, children: Children who receive Busulfan IV and have a pharmacokinetic of Busulfan

SUMMARY:
Test the correlations between the pharmacogenetic and pharmacokinetic of Busulfan IV in children receiving hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Most of the drugs used to treat cancer are metabolized by hepatic enzymes such as cytochrome P450 or Glutathion-S-Transferase (GST). These enzymatic pathways can be more or less active in the drug's metabolism according to the given polymorphism of each patient (pharmacogenomics).

The current hypothesis is that some functional polymorphisms of genes, which control important enzymes in Busulfan metabolism, contribute to the observed interindividual variability in PK of this drug. This variability can hence predict the resistance as well as the toxicity from a drug in patients who have cancer. The pharmacokinetic profile of different drugs, which have a hepatic metabolism, can be dramatically modified by these polymorphisms. Busulfan is a major drug used in the conditioning regimen before hematopoietic stem cell transplantation, particularly in children in whom total body irradiation has to be avoided. This drug has a narrow therapeutic index. At a lower systemic exposure than the targeted one, Busulfan has insufficient activity and hence an increased risk of transplant rejection and leukemic relapse.

At higher systemic exposures, the toxicity risk increases dramatically with an elevated incidence of hepatic veno-occlusive disease (VOD). Pharmacokinetic monitoring of Busulfan allows optimal dosing. The recommended doses are based on the weight, body surface area or age. Nevertheless, a majority of patients will still need an adjustment of the dose administered after their first dose: this will result in a cumulative systemic exposure that will be over or under therapeutic. Busulfan is metabolized principally by the GSTA1, as well as by other GST enzymes like the GSTM1 and GSTP1. These enzymes are present in the liver as well as in the intestinal cells and are up regulated in the digestive system of young children.With this study we will look for the polymorphism in GST genes, look at the Busulfan IV pharmacokinetics and finally look at the GST alpha enzyme activity and see if there is a correlation with clinical end points. This study will also study any correlation with other genes (repair DNA genes, CYP etc..) that could be correlated with Busulfan and/or cyclophosphamide. This study will also allow to do some DNA banking for future studies in genetics. This multicentric study is sponsor by the Swiss pediatric Oncology Group and is a European Bone and Marrow Transplantation study open in 6 countries (Switzerland, Canada, Italy, Holland, Tscèque republic, ). Pilot study are first analyze with St. Justine Hospital then with the other center at a later stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≤ than 18 years of age at study entry on this protocol
* The patient must receive iv Busulfan as part of his hematopoietic stem cell transplant conditioning regimen.
* Each participating center has to go through a PK cross validation
* All patients (or their legal guardians) must sign a document of informed consent that has been approved by the Institutional Human Review Committee.
* Each center has to do his own PK of BU

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: primary care clinic of pediatric
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-02; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
polymorphisms in genes involved in Busulfan pathways correlation with pharmacokinetic | 1 year post hematopoietic stem cell transplantation

SECONDARY OUTCOMES:
polymorphisms in genes involved in Busulfan pathways correlation with toxicity | 1 year post hematopoietic stem cell transplantation
polymorphisms in genes involved in Busulfan pathways correlation with survival | 1 year post stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ansari, MD, PhD, Principal Investigator — Hopital Cantonal de Genève, Switzerland
Locations (4):
- Canada (2):
  - Alberta children's hospital, Calgary, Alberta
  - Chu St Justine, Montreal, Quebec
- Hopital Rebert Debré, Paris, France
- Hopital Cantonal de Genève, Geneva, Switzerland

REFERENCES:
- [Background] Ansari M, Lauzon-Joset JF, Vachon MF, Duval M, Theoret Y, Champagne MA, Krajinovic M. Influence of GST gene polymorphisms on busulfan pharmacokinetics in children. Bone Marrow Transplant. 2010 Feb;45(2):261-7. doi: 10.1038/bmt.2009.143. Epub 2009 Jul 6. PMID 19584821
- [Background] Ansari M, Krajinovic M. Can the pharmacogenetics of GST gene polymorphisms predict the dose of busulfan in pediatric hematopoietic stem cell transplantation? Pharmacogenomics. 2009 Nov;10(11):1729-32. doi: 10.2217/pgs.09.135. No abstract available. PMID 19891548
- [Result] Ansari M, Rezgui MA, Theoret Y, Uppugunduri CR, Mezziani S, Vachon MF, Desjean C, Rousseau J, Labuda M, Przybyla C, Duval M, Champagne M, Peters C, Bittencourt H, Krajinovic M; Pediatric Disease Working Parties of the European Blood and Marrow Transplant Group. Glutathione S-transferase gene variations influence BU pharmacokinetics and outcome of hematopoietic SCT in pediatric patients. Bone Marrow Transplant. 2013 Jul;48(7):939-46. doi: 10.1038/bmt.2012.265. Epub 2013 Jan 7. PMID 23292236
- [Result] Ansari M, Theoret Y, Rezgui MA, Peters C, Mezziani S, Desjean C, Vachon MF, Champagne MA, Duval M, Krajinovic M, Bittencourt H; Pediatric Disease Working Parties of the European Blood and Marrow Transplant Group. Association between busulfan exposure and outcome in children receiving intravenous busulfan before hematopoietic stem cell transplantation. Ther Drug Monit. 2014 Feb;36(1):93-9. doi: 10.1097/FTD.0b013e3182a04fc7. PMID 24061446
- [Result] Huezo-Diaz P, Uppugunduri CR, Tyagi AK, Krajinovic M, Ansari M. Pharmacogenetic aspects of drug metabolizing enzymes in busulfan based conditioning prior to allogenic hematopoietic stem cell transplantation in children. Curr Drug Metab. 2014 Mar;15(3):251-64. doi: 10.2174/1389200215666140202214012. PMID 24524663
- [Result] Uppugunduri CR, Rezgui MA, Diaz PH, Tyagi AK, Rousseau J, Daali Y, Duval M, Bittencourt H, Krajinovic M, Ansari M. The association of cytochrome P450 genetic polymorphisms with sulfolane formation and the efficacy of a busulfan-based conditioning regimen in pediatric patients undergoing hematopoietic stem cell transplantation. Pharmacogenomics J. 2014 Jun;14(3):263-71. doi: 10.1038/tpj.2013.38. Epub 2013 Oct 29. PMID 24165757
- [Result] Acosta-Martin AE, Antinori P, Uppugunduri CRS, Daali Y, Ansari M, Scherl A, Muller M, Lescuyer P. Detection of busulfan adducts on proteins. Rapid Commun Mass Spectrom. 2016 Dec 15;30(23):2517-2528. doi: 10.1002/rcm.7730. PMID 27599297
- [Result] Bartelink IH, Lalmohamed A, van Reij EM, Dvorak CC, Savic RM, Zwaveling J, Bredius RG, Egberts AC, Bierings M, Kletzel M, Shaw PJ, Nath CE, Hempel G, Ansari M, Krajinovic M, Theoret Y, Duval M, Keizer RJ, Bittencourt H, Hassan M, Gungor T, Wynn RF, Veys P, Cuvelier GD, Marktel S, Chiesa R, Cowan MJ, Slatter MA, Stricherz MK, Jennissen C, Long-Boyle JR, Boelens JJ. Association of busulfan exposure with survival and toxicity after haemopoietic cell transplantation in children and young adults: a multicentre, retrospective cohort analysis. Lancet Haematol. 2016 Nov;3(11):e526-e536. doi: 10.1016/S2352-3026(16)30114-4. Epub 2016 Oct 13. PMID 27746112
- [Result] Huezo-Diaz Curtis P, Uppugunduri CRS, Muthukumaran J, Rezgui MA, Peters C, Bader P, Duval M, Bittencourt H, Krajinovic M, Ansari M. Association of CTH variant with sinusoidal obstruction syndrome in children receiving intravenous busulfan and cyclophosphamide before hematopoietic stem cell transplantation. Pharmacogenomics J. 2018 Jan;18(1):64-69. doi: 10.1038/tpj.2016.65. Epub 2016 Oct 25. PMID 27779248
- [Result] Ansari M, Curtis PH, Uppugunduri CRS, Rezgui MA, Nava T, Mlakar V, Lesne L, Theoret Y, Chalandon Y, Dupuis LL, Schechter T, Bartelink IH, Boelens JJ, Bredius R, Dalle JH, Azarnoush S, Sedlacek P, Lewis V, Champagne M, Peters C, Bittencourt H, Krajinovic M. GSTA1 diplotypes affect busulfan clearance and toxicity in children undergoing allogeneic hematopoietic stem cell transplantation: a multicenter study. Oncotarget. 2017 Aug 27;8(53):90852-90867. doi: 10.18632/oncotarget.20310. eCollection 2017 Oct 31. PMID 29207608
- [Derived] Waespe N, Mlakar SJ, Dupanloup I, Rezgui MA, Bittencourt H, Krajinovic M, Kuehni CE, Nava T, Ansari M. A novel integrative multi-omics approach to unravel the genetic determinants of rare diseases with application in sinusoidal obstruction syndrome. PLoS One. 2023 Apr 5;18(4):e0281892. doi: 10.1371/journal.pone.0281892. eCollection 2023. PMID 37018234
- [Derived] Jurkovic Mlakar S, Uppugunduri SCR, Nava T, Mlakar V, Golay H, Robin S, Waespe N, Rezgui MA, Chalandon Y, Boelens JJ, Bredius RGM, Dalle JH, Peters C, Corbacioglu S, Bittencourt H, Krajinovic M, Ansari M; paediatric diseases working party of the European society for blood and marrow transplantation. GSTM1 and GSTT1 double null genotypes determining cell fate and proliferation as potential risk factors of relapse in children with hematological malignancies after hematopoietic stem cell transplantation. J Cancer Res Clin Oncol. 2022 Jan;148(1):71-86. doi: 10.1007/s00432-021-03769-2. Epub 2021 Sep 9. PMID 34499222
- [Derived] Uppugunduri CRS, Storelli F, Mlakar V, Huezo-Diaz Curtis P, Rezgui A, Theoret Y, Marino D, Doffey-Lazeyras F, Chalandon Y, Bader P, Daali Y, Bittencourt H, Krajinovic M, Ansari M. The Association of Combined GSTM1 and CYP2C9 Genotype Status with the Occurrence of Hemorrhagic Cystitis in Pediatric Patients Receiving Myeloablative Conditioning Regimen Prior to Allogeneic Hematopoietic Stem Cell Transplantation. Front Pharmacol. 2017 Jul 11;8:451. doi: 10.3389/fphar.2017.00451. eCollection 2017. PMID 28744217
- See also: European Society for Blood and Marrow Transplantation (EBMT) - Pediatric Diseases Working Party — https://www.ebmt.org/working-parties/paediatric-diseases-working-party-pdwp